CLINICAL TRIAL: NCT02452957
Title: A Prospective Multi-Center Study of the Safety and Effectiveness of the Tornier Simpliciti™ Shoulder System in Shoulder Arthroplasty
Brief Title: Safety and Effectiveness of the Tornier Simpliciti™ Shoulder System in Shoulder Arthroplasty
Status: Withdrawn | Type: Observational
Why Stopped: Contract issues
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: 1206-T-SIMPLICITI-RM
Record Dates: First submitted 2015-05-16; First posted 2015-05-25 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-03

CONDITIONS: Shoulder Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Device: Simpliciti™ System: The Simpliciti™ nucleus is a humeral prosthesis intended for total and hemi shoulder arthroplasty in patients with a severely painful and/or disabled joint resulting from osteoarthritis or traumatic arthritis.
  The implant is sized to match and replicate the anatomy of the proximal humerus, while maintaining a bone conserving approach. It does not extend beyond the metaphysis, leaving the humeral canal untouched. Fixation is enhanced through a porous coating with a high coefficient of friction; resulting in a solid initial fit and long term fixation.
  The Simpliciti™ nucleus is designed to receive a humeral head. The Simpliciti™ system is authorized to bear the CE mark and will be investigated within this clinical study in accordance with its intended use.

SUMMARY:
The aim of this observationnal post-marketing study is to provide additional information on the safety and effectiveness of Simpliciti™ system at 24 months post-shoulder arthroplasty , in usual surgical practice.

ELIGIBILITY:
Inclusion Criteria:

* A subject must meet all of the following inclusion criteria in order to enter the study:

  * Adult subject 18 years or older,
  * Clinical indication for total shoulder or hemi replacement due to primary diagnosis of osteoarthritis,
  * Scapula and proximal humerus must have reached skeletal maturity,
  * Willing and able to comply with the protocol,
  * Willing and able to personally sign the informed consent form,
  * Subject is legally competent, understands the nature, significance and implications of the clinical investigation, and is able to form a rational intention in the light of these facts.

Exclusion Criteria:

* A subject will not be eligible to participate in the study if any of the following conditions is present:

  * lack of sufficient sound bone to seat and support the implant, including that resulting from skeletal immaturity, osteoporosis or erosive arthritis,
  * Severe Walch grade B2 glenoid defined as >60% posterior head displacement and >20% posterior glenoid bone loss,
  * metal allergies or sensitivity,
  * infection at or near the site of implantation,
  * distant or systemic infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subject with clinical indication for total shoulder or hemi replacement due to primary diagnosis of osteoarthritis.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with device related adverse events as a measure of safety | 24 months
  All adverse events will be summarized by the number and percentage of patients with each type of event. The following will be summarized separately: procedure related adverse events, device related adverse events, anticipated adverse events. Additionally, the incidence of serious device associated adverse events will be summarized.

SECONDARY OUTCOMES:
Change in the Range of Motions (ROM) as a measure of effectiveness | 24 months
  Changes in ROM variables from the pre-implant visit to each follow-up visit will be calculated and sumarized until 24-month visit.
Change in the Constant Score as a measure of effectiveness | 24 months
  Changes in the Constant Score from the pre-implant visit to each follow-up visits will be calculated and summarized until 24-month visit.
Change in the DASH Score as a measure of improvement in the patients' Quality of Life | 24 months
  Changes in the DASH Score from the pre-implant visit to each follow-up visits will be calculated and summarised until 24-month visit.
Change in humeral cortical thickness as an evaluation of Stress Shielding | 24 months
  Changes in humeral cortical thickness from the pre-implant to 24-month visit will be mesured according to the modified method of Tingart & Al.

CONTACTS AND LOCATIONS:
Overall Officials: Steve A. Erickson, Study Director — Stryker Trauma and Extremities; Ulrich Brunner, MD, Prof., Principal Investigator — Krankenhaus Agatharied
Locations (1):
- Krankenhaus Agatharied, Hausham, Germany